CLINICAL TRIAL: NCT04571788
Title: Treating Rhegmatogenous Retinal Detachment by Foldable Capsular Buckle (FCB): a Randomized, Controlled, Single-blind and Multicenter Study
Brief Title: Treating Rhegmatogenous Retinal Detachment by Foldable Capsular Buckle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: AIER2019IRB10
Record Dates: First submitted 2020-09-06; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Rhegmatogenous Retinal Detachment; Surgery
Keywords: Rhegmatogenous Retinal Detachment; Foldable Capsular Buckle; Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FCB group: FCB group received FCB implantation
  Interventions: Procedure: Foldable Capsular Buckle
- Control group: Control group undergoes silicone scleral pad surgery
  Interventions: Procedure: Silicone scleral padding

INTERVENTIONS:
Procedure: Foldable Capsular Buckle — Intraoperatively, the location and size of the fissure hole is located under the microscope to determine the location and extent of the conjunctival incision. Once local infiltration anesthesia is complete, a 2 ml needle is inserted into the outer surface of the sclera >10 mm behind the corneoscleral rim, and a cotton swab is used to apply light pressure on the side of the wound to help drain the fluid. Under the microscope, the emptied and folded FCB was inserted vertically into the external scleral channel and the drainage valve was sutured with 5.0 non-absorbable sutures 8-10 mm behind the angular scleral rim. The balloon was then filled with 1 ml of alkaline Ringer's solution using a 1 ml syringe through the drainage valve. Subconjunctival injection of tobramycin and dexamethasone was followed by gentle pressure and bandaging of the eye.
  Groups: FCB group
Procedure: Silicone scleral padding — Intraoperatively, the location and size of the fissure is located under the microscope to determine the location and extent of the incision of the bulbar conjunctiva. When the fissure hole is located microscopically, a retrobulbar block anesthesia is performed and fluid is released according to the degree of retinal detachment. Silicone was then implanted on the scleral surface as an external cushion and intraocular pressure was applied, and the opening was finally sutured, with laser closure performed within a week after surgery. After the surgery, subconjunctival injection of tobramycin and dexamethasone was routinely performed, and the operated eye was bandaged, with observation of the fundus and closure of the aperture.
  Groups: Control group

SUMMARY:
To evaluate the efﬁcacy and safety of treating rhegmatogenous retinal detachment (RRD) using foldable capsular buckle (FCB). It is a multi-center clinical ,randomized, controlled, and single-blind clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety, effectiveness, and operability of FCB scleral buckling and silicone scleral buckling in the treatment of RRD. It is a multi-center clinical study and is designed according to a randomized, controlled, and single-blind clinical research protocol. Before surgery, the retinal tear in the FCB group and the control group of RRD patients should be examined and precise positioned by fundus photography, and the relevant results will be determined by the third-party reading center to confirm that the patients can accept such surgery.

The key instrument required by the FCB group is FCB. During FCB implantation, 1 ml of basic Ringer's solution will be injected as FCB, and then the balloon filled, so that the outer surface of the balloon is in close contact with the sclera, and the top The function of scleral compression helps to close the hiatus. The key surgical instrument used in the control group is silicone, but it does not require ring surgery. Silicone is also fixed to the outer surface of the sclera. After the conjunctiva and Tenon 's sac separated, the primary endpoint will be evaluated three months after surgery, and both groups will be followed up to one year after surgery. Relevant data will be collected and kept by full-time personnel, and then the statistical analysis of the data will be used to evaluate the safety, effectiveness, and operability of FCB implantation, and compare the treatment effect with the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, regardless of gender.
* The axial length of the operative eye ≤26 mm (myopia <600 degrees).
* Meet diagnostic criteria for RRD (a single lacuna of <2 PD in one quadrant or multiple adjacent lacunae of <3 PD, up to PVR-B grade).
* Be able to understand the purpose of the study, participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* Patients with known allergies to silicone, scarred bodies.
* Intraocular inflammation.
* PVR-C and above.
* Cracked hole with crimped edges, with pulling.
* Obvious vitreous pulling and retinal fixation folds.
* the lacunae are large or scattered and the scleral ridge formed by the estimated FCB does not fully encompass the lacunae.
* Other associated ophthalmic diseases beyond control, such as glaucoma, tertiary nuclear cataracts and macular diseases.
* Severe hepatic and renal impairment and/or severe systemic diseases (e.g. cardiovascular, respiratory, digestive, neurological, endocrine, genitourinary, etc.).
* Females who are already pregnant (determined by urine pregnancy study at the first visit), who are preparing for pregnancy during the study and who are lactating.
* History of substance abuse or alcoholism.
* Have participated in another clinical study of a drug or medical device within 30 days prior to the screening of this clinical study.
* Any condition of the patient that the research doctor believes would hinder clinical research (e.g. the patient is prone to stress, uncontrolled emotions, depression, etc.).
* Those who do not agree to be selected or do not agree to be followed up.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who meet the diagnostic criteria for RRD (single fissure in one quadrant of <2 PD or adjacent multiple fissures of <3 PD, below PVR-B grade).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
fundus photography | 12 weeks after surgery
  The retinal repositioning will be observed and the images will be reviewed by a third-party film review committee for final results.
Optical Coherence Tomography, OCT | 24 weeks after surgery
  Check to see if the retina is reset.The macula is defined as a central depression within a diameter of 5.5 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Shibo Tang, Prof, Principal Investigator — Aier School of Ophthalmology, Central South University
Locations (1):
- Aier School of Ophthalmology, Central South University, Changsha, Hunan, China